CLINICAL TRIAL: NCT00591877
Title: A Study to Evaluate the Role of Alternative Medicine in Difficult to Treat GERD Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll elegible subjects. No subjects enrolled, study closed.
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, PRATEEK SHARMA, Principal Investigator, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PS0045
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERDCAM: Complementary and alternative medicine; NERD: non-erosive reflux disease; GERD: gastroesophageal reflux disease; AC: acupuncture; SAC: sham acupuncture; LES: lower esophageal sphincter pressure; TLESR: transient lower esophageal sphincter relaxation; Acupuncture; Yoga
MeSH Terms: conditions — Gastroesophageal Reflux; Non-Erosive Reflux Disease | interventions — Acupuncture Therapy; Yoga

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AC (Active Comparator): Acupuncture:
  The patients will receive acupuncture by a trained doctor with acupuncture expertise, at 3 points relevant to reflux symptoms. Each patient will undergo a 30 minute session, twice a week, for a total of 12 sessions. The technique will involve electro-stimulation at predefined points followed by needle manipulation.
  Interventions: Procedure: Acupuncture
- SAC (Sham Comparator): The patients randomized to this arm will receive acupuncture for a similar duration and number of sessions. The sham acupoints are at least 2 cm away from the actual acupoints to prevent acupressure effects
  Interventions: Procedure: Sham Acupuncture
- Yoga (Active Comparator): The participants in this arm will undergo a 60 min session of yoga exercises. These exercises are specifically designed for reflux symptoms by a yoga instructor. This includes a set of specific physical postures (asana) and breathing techniques within the four-element setup. The set of asana are divided into (a) standing, (b) sitting, and (c) lying down positions. The session will begin with asana in standing position, followed by a position called Shavasan (relaxation), then asana in sitting down position followed by Shavasan, finally asana in lying down position followed by Shavasan. At the end of all asana, Pranayam (special breathing exercises) will be practiced.
  Interventions: Other: Yoga

INTERVENTIONS:
Procedure: Acupuncture — Each patient will undergo a 30 minute session, twice a week, for a total of 12 sessions. The technique will involve electro-stimulation at predefined points followed by needle manipulation.
  The acupoints that will be used are:
  * ST-36: 3 finger breadths inferior to lower edge of patella between tibialis anterior muscle and the tibia, 1 finger breadth lateral to the anterior crest of the tibia.
  * PC-6: 2 finger breadths proximal to and in the middle of the most distal transverse crease of the wrist, between the tendons of palmaris longus and flexor carpi radialis.
  * CV-12: 4 finger breadths superior to the umbilicus.
  Other Names: AC
  Arms: AC
Procedure: Sham Acupuncture — The acupoints for SAC are:
  * LI-4 : adjacent to and at the middle of the radial side of the 2nd metacarpal bone, at the same level as the end of the crease when the thumb and index fingers approximate.
  * GB-32: on the lateral aspect of the thigh 5 finger breadths proximal to the popliteal crease, 2 finger breadths inferior to GB31.
  * UB -15: 1.5 finger breadths lateral to the midline of the spine on a level between the 5 th and the 6 th thoracic vertebrae.
  Other Names: SAC
  Arms: SAC
Other: Yoga — The participants in this arm will undergo a 60 min session of yoga exercises. These exercises are specifically designed for reflux symptoms by a yoga instructor. This includes a set of specific physical postures (asana) and breathing techniques within the four-element setup. The set of asana are divided into (a) standing, (b) sitting, and (c) lying down positions. The session will begin with asana in standing position, followed by a position called Shavasan (relaxation), then asana in sitting down position followed by Shavasan, finally asana in lying down position followed by Shavasan. At the end of all asana, Pranayam (special breathing exercises) will be practiced.
  Arms: Yoga

SUMMARY:
Patients with refractory GERD on BID PPI's assigned to the acupuncture group will have significant improvement in their symptoms after receiving acupuncture for 6 weeks as compared to sham acupuncture given for the same duration.

Primary Aim 1:To determine the efficacy of acupuncture in the treatment of refractory GERD.

Participants with refractory GERD on BID PPIs randomized to yoga will have a significant relief in the symptoms of reflux.

Primary Aim 2:To determine the efficacy of yoga in the treatment of refractory GERD.

DETAILED DESCRIPTION:
BACKGROUND

Prevalence and burden of disease:

Gastroesophageal reflux disease (GERD) defined as presence of symptoms of heartburn and/or acid regurgitation is a common chronic disorder. It is a significant health problem especially in the Western population associated with a huge economic burden and impaired quality of life (1, 2). The prevalence of GERD in the adult population of the United States is 40% (symptoms at least once a month). Approximately 20% report GERD related symptoms weekly while 14% report them on a daily basis.

The leading gastrointestinal symptoms evaluated in a primary care office setting are those related to a diagnosis of GERD. The mainstay of treatment for GERD symptoms at present time are proton pump inhibitors (PPI) in combination with life style changes. In fact, PPI have become one of the most commonly written prescriptions, trends suggesting that per year scripts have doubled since 1999. It is estimated that Americans spend in excess of 10 billion US dollars/year on PPIs and two of the top five selling drugs in the United States are PPIs (5). For patients who prefer to refrain from long-term medication use, may benefit from acid-reflux surgeries such as Nissen fundoplication. However, acid-reflux reducing procedures are associated with operative morbidity and mortality including several complications including gas bloat syndrome. A large number of patients who undergo surgery for reflux symptoms may eventually relapse and require PPIs. Thus, treatment of reflux, either pharmacological or surgical, is costly (6-9) and presents a significant economic burden on the health-care delivery system.

Social Impact of the disease:

GERD symptoms are associated with bodily pain, impaired social, emotional and physical functioning which has a profound impact on daily living. Much research has been done to evaluate the true burden of GERD on our society. For instance, 40% of patients with nighttime symptoms of GERD reported that such symptoms affected their ability to function the next day. Furthermore, 27% of these patients reported that their own night-time symptoms affected their spouses ability to sleep (10). Clearly, this data indicates a huge number of Americans who report the effects of heartburn on personal and spousal quality of life. GERD symptoms need to be addressed effectively as successful treatment for GERD results in improvements in health related quality of life (11, 12). In the treatment of GERD, the goal should be complete symptom resolution as this has been shown to be associated with a clinically significant improvement in health related quality of life (HRQL) (13).

Refractory GERD:

Despite life style changes and compliant therapy with PPI, a large number of patients may have persistent symptoms and classified to have refractory GERD, a distinctive group that is difficult to manage (14). The putative reasons remain poorly defined but likely include contributions from factors such as non-acid reflux, visceral hypersensitivity, and abnormal esophageal motor events (14). A study by Tack et al investigated mechanisms for poor response to PPI therapy and showed persistence of acid reflux in 11%, bile reflux alone in 38% and a combination of acid and bile reflux in 26%. However, persistence of acid or bile reflux does not prove a causal relationship with symptoms (15). Also, in this group of individuals with acid or bile reflux on BID PPI's, a possible treatment option is Nissen's fundoplication, the utility of which is yet to be proven in this cohort. There is no consensus definition of refractory GERD and generally, it is defined as non-response of symptoms to optimum PPI trial. The goal of providing symptomatic relief to these refractory patients is extremely challenging in view of limited options. It is to these patients that the investigators would like to evaluate in a feasibility study the use of complementary medicine modalities including acupuncture and yoga that may be relatively safe, cost-effective therapies to help with the distressing symptoms of GERD.

Complementary and alternative medicine:

Complementary and alternative medicine (CAM) is a group of diverse medical and health care systems, therapies and products that are not presently considered to be part of conventional medicine. These methods have been used for centuries in the eastern culture for a myriad group of diseases. CAM became popular in the US in the 1990's where majority of people used it as a complement to conventional medicine and not as an alternative (16-18). Recently, there has been much interest in applying these modalities not as secondary therapies to conventional treatment but as the primary method. Amongst them acupuncture and yoga have gained a great deal of popularity.

Acupuncture (AC):

Acupuncture is part of the traditional Chinese medicine a complete system of healing that dates back to 200 BC. The general theory of acupuncture is based on the premise that there are patterns of energy flow (Qi) through the body that are essential for health and disruptions of this flow are believed to be responsible for disease. Studies have shown that AC modulates the endorphin system via the central pain processing pathways (19, 20). Acupuncture has been widely used for various gastrointestinal disorders. It is conceivable that acupuncture may be effective in patients with GERD because it has been shown to alter acid secretion, GI motility and visceral pain (21, 22).

The pathogenesis of GERD is multifactorial. The predominant mechanism postulated to cause GERD is transient relaxation of the lower esophageal sphincter (TLESR). Pathological reflux may also occur due to low LES pressures (23). Studies have shown that acupoint stimulation can decrease the rate of TLESR's and hence prevents reflux (24). The investigators propose to use 3 acupoints ST-36, PC-6, CV-12 for treatment of symptoms of GERD. These points are described in the subsequent sections. Acupuncture will be performed by Dr. Santosh Sharma who has the expertise in this treatment modality and is currently offering his therapy for several years at the Veterans Affairs Medical Center, Kansas City.

Yoga:

Yoga refers to a combination of breathing exercises and postures designed to involve specific muscle groups with systemic effects on the various organ systems. Yoga originated in India at least 3000 years ago. The practice of yoga came to US in 1890 and gained popularity in 1960s because of a rising interest in and cultural acceptance of alternative modalities and mind body therapies. Yoga is offered in local YWCA, health clubs and yoga centers and in hospitals as part of disease prevention and management programs (25).The most popular form is Hatha yoga. As discussed below, the usefulness of yoga has been studied in certain chronic illnesses such as back pain with promising results. The investigators propose to use yoga exercises specifically designed for reflux symptoms. Dr. Vijay Kumar will be offering yoga classes to patients with refractory GERD. Dr. Vijay Kumar is a Professor of Computer Science at University of Missouri - Kansas City and has been offering classes for several years at various levels.

Evidence for use of acupuncture and yoga:

Several randomized controlled trials have been conducted demonstrating the beneficial effects of acupuncture. A randomized controlled study in 29 patients with mild to moderate ulcerative colitis with a 4 month follow up after completion of acupuncture sessions showed a statistically significant improvement in colitis activity index (CAI) as compared to the control group. The study concluded that acupuncture provided an additional therapeutic benefit to patients with mild to moderate ulcerative colitis (26).

Another randomized 3-arm study was conducted to assess the efficacy and safety of traditional Chinese acupuncture compared with sham acupuncture (needling at defined non-acupuncture points) and conservative therapy in patients with chronic pain due to osteoarthritis of the knee. Addition of acupuncture led to significant improvement in the symptoms (27). Recently, Dickman et al evaluated the efficacy of adding acupuncture (twice a week over 4 weeks) as compared to doubling the PPI dose in 30 refractory GERD patients(28). The acupuncture group demonstrated a significant decrease in mean daytime heartburn scores compared to high-dose PPI group. Mean nighttime heartburn and regurgitation scores improved only in the acupuncture group. Thus this study showed that adding acupuncture as compared to doubling the PPI dose was more effective in controlling symptoms of GERD in patients on standard dose of PPI.

Similar benefits have been demonstrated with the use of yoga. A randomized controlled trial compared yoga, exercise and self care book for chronic low back pain showed that yoga was more effective than a self-care book for improving function and reducing chronic low back pain and the benefits persisted for at least several months (29). Yoga was also found to be useful in improving symptoms related to irritable bowel in a randomized trial conducted in Canada (30).

CLINICAL RELEVANCE OF THIS STUDY GERD is a well known, widely prevalent, clinical entity. The symptoms of GERD if not relieved can affect the daily functioning/productivity of individuals. This can be especially frustrating for some patients, who may spend hundreds of dollars every year on prescription medications, and are still not able to obtain relief of their symptoms. In the United States alone, it is estimated that PPI costs alone make up over $10billion/year (5). However, despite these staggering costs, it is clear that even PPI therapy is not the definitive answer for all patients. Indeed, it has been reported that 37% of patients receiving PPIs also note concomitant antacid use. This finding underscores the fact that even with PPI therapy, a large percentage of patients do not achieve full symptom relief. When left untreated--or when treated inadequately--severe GERD can progress to esophagitis, esophageal ulcers, esophageal strictures, laryngeal disease, chronic cough, Barrett's esophagus, and esophageal adenocarcinoma. Clearly, such patients with refractory symptoms are the ones in the direst need for additional modalities of therapy. Yoga and acupuncture may be a promising option for these patients, as they represent cost-effective, yet underused, options which may be usefully employed to control the symptoms of GERD.

Data Collection:

Patient demographics, order of randomization, responses to questionnaires, and antacid use will be collected by the study coordinator and recorded in a database.

RISK AND BENEFIT TO THE STUDY PARTICIPANT:

This pilot prospective study has the potential to identify new treatments for GERD symptoms. The participants in this study may experience relief from their GERD symptoms persistent on high dose acid suppressive therapy. This may improve their quality of life and level of functioning. The risks to the study group are minimal. There is minor risk of bruising, needle breakage and infection with the acupuncture needles and musculoskeletal symptoms in patients undergoing yoga. If the study shows significant improvement in reflux symptoms with acupuncture or yoga, then these methods may have a wider application to the entire spectrum of GERD symptoms with the prospect of avoiding pharmacologic and surgical therapies.

STATISTICAL METHODS AND DATA ANALYSIS:

Data Analysis:

Data will be analyzed with the help of a statistical software program. Categorical and continuous variables will be compared using the Student's t-test and chi-square test. A p value of < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be a Kansas City VA Hospital patient.
* 18 yrs or older.
* agreeable to randomization.
* patients with refractory GERD on bid PPI.
* negative endoscopy in the last 5 yrs.
* able to follow simple instructions and perform simple exercises.
* capable of giving informed consent.

Exclusion Criteria:

* GERD with known complications e.g. peptic stricture.
* Hepatitis C.
* HIV.
* Peripheral neuropathy.
* Irritable bowel syndrome
* Previous acupuncture.
* any other major co morbidity e.g. scleroderma etc.
* chronic anticoagulation.
* pregnancy/lactation.
* prior h/o esophageal surgery.
* H/o of Barrett's esophagus.
* Esophageal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Decrease by 50% in the RDQ scores as compared to baseline at the end of the study period | 1 year

SECONDARY OUTCOMES:
Improvement in reflux related quality of life (QOLRAD) scores at the end of the study by 50% | 1 year
Decrease by 50% in the baseline RDQ scores at 12 and 26 week follow up after the completion of the study | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Kansas City VA Medical Center
Locations (1):
- Kansas city VA Medical center, Kansas City, Missouri, United States